CLINICAL TRIAL: NCT05721170
Title: Impact of Beta-blockers Among Patients Undergoing TAVI: a Randomized Multicenter Trial
Brief Title: Impact of Beta Blockers on TAVI (BETA-TAVI)
Acronym: BETA-TAVI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Professor of Cardiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BETA-TAVI Trial
Record Dates: First submitted 2023-01-28; First posted 2023-02-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; Aortic valve stenosis; TAVR; Pacemaker implantation; Beta blocker
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Intervention Model Description: Eligible patients will be assigned randomly in 1:1 ratio to either continue or withdraw the already receiving beta-blockers medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-blockers continuation (Active Comparator): Patients assigned in the beta-blockers continuation arm will be receiving per os beta blocker medication for at least 72 hours before TAVI without interruption after it.
  Interventions: Drug: Beta blocker
- Beta-blockers interruption (Active Comparator): Patients assigned to interrupt the beta-blockers treatment will abstain from beta blockers for at least 7 days after TAVI.
  Interventions: Drug: Beta blocker

INTERVENTIONS:
Drug: Beta blocker — Investigation on beta-blockers in TAVI and brief post-TAVI period.

SUMMARY:
This is a prospective, multicentre, investigator-initiated, randomized clinical trial clinical trial investigating the impact of beta-blockers administration among patients undergoing TAVI for severe aortic valve stenosis. Adults already receiving beta-blockers be assigned randomly in 1:1 ratio to either continue or withdraw the beta-blockers medication at least 72 hours before and at least 7 days after TAVI. The primary endpoint is permanent pacemaker implantation rates in 7 days after the procedure. Secondary endpoints include death, cardiogenic shock and arrhythmias/conduction abmormalities with time frame 12 months.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE Aortic Stenosis is the most common valvulopathy in the developed world. Approximately, 5% of people over 65 years old, in the general population, suffer from aortic stenosis, and the percentage increases with aging. The natural progress of the disease consists of a long-term asymptomatic period with low morbidity and mortality, followed by the symptomatic period. However, the symptoms manifestation (such as syncope, angina, dyspnea and heart failure) is accompanied by a serious increase in morbidity and mortality. The standard diagnostic technique is the transthoracic cardiac ultrasound. Transcatheter aortic valve implantation (TAVI) is an established and valuable treatment option for patients with both severe symptomatic aortic stenosis and increased risk for surgical aortic valve replacement (SAVR). The use of TAVI is rapidly expanding worldwide and the indications are widening into lower-risk populations in view of favorable outcomes among high and intermediate-risk patients.

   Treatment with beta-blockers is a cornerstone for patients belonging to the wide range of heart failure, especially in those with heart failure with reduced ejection fraction. They are also widely used for the management of various arrhythmias and sudden cardiac death prevention as well as coronary artery disease. Severe valvulopathy is a major cause of heart failure and arrhythmogenesis but the role of beta-blockers in the valvulopathies per se is not clarified.

   Increased left ventricular intracavital gradient leading to mid-ventricular or outflow tract obstruction with potentially severe hemodynamic compromise has been described in patients with left ventricular hypertrophy undergoing SAVR. The term "suicide left ventricle" has been adopted for this clinical setting and is possible to be revealed after TAVI as well. Beta-blocker administration is a recognized way to alleviate left ventricular outflow tract (LVOT) obstruction in patients with obstructive hypertrophic cardiomyopathy and may also prevent or decrease intracavital gradients after TAVI. However, as a way to avoid conduction abnormalities and permanent pacemaker implantation (PPI) after TAVI, it is common for operators to withdraw beta-blockers before TAVI.

   A large observational trial from the OCEAN-TAVI registry comparing with propensity-matching patients undergoing TAVI with or without beta-blockers exhibited no significant differences in PPI between the two groups. Another observational trial investigating arrhythmic risk in TAVI patients regarding beta-blocker administration concluded that beta-blocker withdrawal was associated with increased arrhythmic burden and more PPIs. The latter paradoxical outcome was attributed by the authors to sick sinus syndrome revelation secondary to increased atrial fibrillation (AF) development in patients who discontinued beta-blockers.

   Clinical data concerning this topic are scarce and the safety and efficiency of beta-blockers during and post-TAVI are not well-documented. The aim of this clinical trial is to investigate the impact of beta-blocker administration among patients undergoing TAVI.
2. DESCRIPTION OF THE PROTOCOL 2.1 Study design This a prospective, multicentre, investigator-initiated, randomized clinical trial investigating the impact of beta-blockers administration among patients undergoing TAVI.

   2.2 Study population Eligible patients are adults that whom TAVI is indicated as therapy for severe aortic valve stenosis and will be assigned randomly in a 1:1 ratio to either continue or withdraw the beta-blockers medication. Furthermore, they should satisfy all eligibility criteria (inclusion and exclusion).

   2.3 Study centers Hospitals with operators experienced in TAVI operations will be selected. 2.4 Study period This study is expected to be initiated in June 2024. The end of the study is 12 months after the enrollment of the last patient.

   2.5 Informed consent Enrolment can be started when signed informed consent has been obtained. The investigator will explain the nature of the inventory, potential risks and benefits of participation, and answer questions for the patient. All patients must provide informed consent in accordance with the local Institutional Review Board (IRB), using an IRB-approved informed consent form. Any of the patients, who already provided informed consent to this trial, can withdraw their consent from the study any time.
3. STUDY PROCEDURES 3.1 Pre-procedure Screening visit Patients potentially eligible for the BETA-TAVI trial may be screened up to 3 months before TAVI. Medical history and medication will be obtained and clinical examination, ECG, transthoracic cardiac ultrasound (TTE) and blood tests (Appendix) will be performed. Based on the above screening for eligibility criteria will be made.

   Randomization visit Randomization will be performed in a 1:1 ratio, with asymptotic maximal method and maximally tolerated imbalance 3. The National Cancer Institute Clinical Trial Randomization tool will be used. The principal researchers will remain blinded to the allocation sequence to eliminate selection bias. The randomized results will be restricted to a third party who will reveal each successive trial's participant allocation only after that participant has been accepted into the trial.

   Patients eligible for enrolment (every inclusion and no exclusion criteria should be met) may be randomized at least at 72 hours before TAVI. Patient preparation will take place in accordance with standard hospital policy for the care of patients undergoing TAVI. Patients assigned in the beta-blockers continuation arm will be receiving per os beta-blocker medication (the same active pharmaceutical substance) for at least 72 hours before TAVI without interruption after it. Patients assigned to interrupt the beta-blockers treatment will abstain from beta-blockers for 72 hours before TAVI.

   3.2 Medication Patients will receive appropriate antithrombotic and antibiotic medication according to standard hospital and operators' practice.

   3.3 TAVI procedure Qualifying subjects will undergo TAVI procedure. The access site and the prosthetic valve type and size will be selected by the operators. The necessity of balloon pre and/or post-dilatation will be at the discretion of each operator. The type of anesthesia (local, general, sedation) will be selected by the operators as well. Every step and complication that occurred and materials and techniques that were used will be cataloged.

   3.4 Post-procedural care Following the procedure, the patient will be treated in accordance with hospital standard of care. ECG and laboratory blood tests (Appendix) will be obtained post-TAVI and during hospitalization as necessary. A Post-TAVI TTE will be performed as well. Any possible complication or adverse event will be managed based on the nature of the event according to local policy. In the interruption arm, beta-blockers could be reinitiated the sooner 7 days after TAVI. Patients belonging to the continuation arm should continue treatment for at least 7 days after TAVI. Efforts will be made to adhere to the protocol; however, patients' safety is prioritized and in case of adverse events or endpoints that require immediate initiation or interruption of beta-blockers the attending physicians may proceed to interruption or initiation of beta-blockers medication. In that case the endpoint(s) will be cataloged and the patient will continue the participation in the trial adhering to the modified beta-clocker treatment (crossover). Any dose modification will be cataloged as well.

   3.5 Follow-up Follow-up examination will be performed in discharge, 7 days, 30 days and 12 months. At the visits, any adverse event or endpoint will be cataloged. ECG, TTE and laboratory tests will be part of the visit.
4. ENDPOINT MEASURES 4.1 Primary endpoint The trial's primary endpoint is PPI rates (time frame: 7 days). The indications of PPI are mentioned in the 2021 European Society of Cardiology Guidelines on cardiac pacing and cardiac resynchronization therapy.

   4.2 Secondary endpoints
   * All-cause mortality (time frame: 12 months).
   * Cardiovascular mortality (time frame: 12 months).
   * PPI rates (time frame 7days to 12months).
   * Shock needing inotropic or vasoconstrictive medication (time frame: 12 months).
   * New documented atrial fibrillation/flutter (time frame: 12 months).
   * New documented ventricular tachycardia/fibrillation (time frame: 12 months).
   * New RBBB (time frame: 12 months).
   * New LBBB (time frame: 12 months).
   * New 1st degree AV block (time frame: 12 months).
   * New severe bradycardia (<50 beats per minute) (time frame: 12 months).
5. SUBJECT SAFETY This trial intends to clarify the role and impact of beta-blockers in TAVI procedures. This single intervention could provide hemodynamic benefits to the patient, whereas from the available clinical data, no increased risk of PPI is documented. The procedural screening, preparation and the procedure itself of the patients will not be affected by this study. The standard TAVI (in patients without an implanted permanent pacemaker) is being performed with a temporary pacemaker electrode in the right ventricle to enable rapid ventricular pacing and as a backup in case of high-degree conduction abnormalities and bradycardia. This step ensures the patient's safety in the case of beta-blocker contribution to the conduction abnormalities or bradycardia. The thorough monitoring of the patients during TAVI and hospitalization further increases safety. Beta-blockers will be only received by patients for whom there is an indication according to international guidelines. Heart failure with reduced or mildly reduced ejection fraction, atrial fibrillation, atrial or ventricular arrhythmogenesis, symptomatic stable coronary artery disease and prior myocardial infarction are the most frequently encountered diseases that beta-blockers are indicated.
6. STATISTICAL CONSIDERATIONS 6.1 Sample size The incidence of PPI (primary endpoint) was calculated at 12.4% for patients under beta-blockers and 11.3% for patients in a primary observational trial by Saito et al.(16). As 11.3% was the point estimate, the steering committee of the BETA-TAVI trial considered that beta-blocker administration for TAVI could be regarded as non-inferior to no beta-blocker in the lower margin of the confidence interval does not lie above the rate of 11.3% by more than 8% (i.e., if it is not >19.3%). Based on these assumptions, we expect that a sample size of 312 patients is required to achieve 80% power to demonstrate the safety of beta-blockers administration when the type I error rate is set at 0.05. To eliminate the possible impact of a small dropout rate of 10%, we aimed to recruit a total of 347 patients.

   6.2 Statistical analysis All safety and efficacy outcomes will be summarized using descriptive statistics. All patients who have been randomized to study treatment will be included in analysis irrespective of their protocol adherence and continued participation in the study. The primary analysis will be based on the intention to treat (ITT) principle using events confirmed by adjudication.

   6.3 Subgroup prespecified analysis Analyses involving multivariate analysis will be used to evaluate the primary outcome incidence in the prespecified subgroup (section 3.3).
7. ETHICAL AND REGULATORY STANDARDS This study complies with the principles laid down by the 18th World Medical Assembly (Helsinki, 1964) and all applicable amendments laid down by the World Medical Assemblies, and the ICH and GCP guidelines. The local IRB has approved the realization of this trial (General Hospital of Athens "Hippokration" IRB decision No19 of 26th/13Dec2022 meeting with protocol number 22271-27/12/2022).

   7.1 Privacy protection Subjects participating in this study will be given a specific code. There will be no patients' information, which can be utilized to identify patients, stored in the e-CRF. Data that are being stored such as year of birth, date of examination, and age /sex of the subject amongst other things, but none of which will identify the specific subject. Although Ethical Committee may examine adverse event form, case report form and so on during or after clinical trial, no identifiable data will be provided even in this case. In case identification of a specific subject is needed, one needs to obtain access to the hospital records which are already protected.

   This study does not involve the obtaining or inclusion of body material. In case during the study an unexpected finding is obtained concerning the health of the involved subject. The subject involved will be informed at the time of test. If the subject does not wish to be informed then he/she will not be able to participate in this study. Subjects are allowed to withdraw from this study at any time. Information gathered, however, will be used where applicable for the results of the study.

   7.2 Conflict of interest No conflict of interest is present. 7.3 Informed consent The investigator, or a person designated by the investigator, should fully inform the subject of all pertinent aspects of the clinical study including the written information given approval / favorable opinion by the Ethics Committee or the institution's appropriate scientific board (IRB). Prior to a subject's participation in the clinical study, the Informed Consent Form should be signed and personally dated by the subject and by the person who conducted the informed consent discussion.
8. STUDY MONITORING 8.1 Responsibility of the Investigators The investigators undertake to perform the study in accordance with this protocol and Good Clinical Practice. For the trial duration, the investigator(s) will maintain complete and accurate documentation including - but not limited to - medical records, trial progress records, laboratory reports, case report forms, signed informed consent forms, device accountability records, correspondence with the IRB, adverse event reports, and information regarding patient discontinuation or completion of the trial.

   8.2 Case Report forms It is the responsibility of the investigator to maintain an accurate e-CRF to record all observations and other data pertinent to the clinical and laboratory investigations. All e-CRFs should be completed in their entirety in a neat, legible manner to ensure accurate interpretation of data. The data may be recorded either on hard copies (case report forms) or electronic data capture. This data will be monitored by and forwarded to the PI in an expedited fashion.
9. ADVERSE EVENTS All events will be registered in the e-CRF. Adverse events will be actively checked during follow-up. The patient folder will provide contact information for patients in case of questions and when complications occur.
10. PUBLIC DISCLOSURE AND PUBLICATION POLICY Regardless of the results of this study maximum effort for publication will be made.
11. RECORD RETENTION The investigator(s) will maintain all records pertaining to this study for fifteen years after the study is discontinued.

ELIGIBILITY:
Study population

Eligible patients are adults that whom TAVI is indicated as therapy for severe aortic valve stenosis and will be assigned randomly in a 1:1 ratio to either continue or withdraw the beta-blockers medication. Furthermore, they should satisfy all eligibility criteria (inclusion and exclusion).

Inclusion criteria

* Adults ≥18 years old.
* Patient with severe symptomatic aortic stenosis defined by mean aortic gradient > 40 mmHg or/and peak jet velocity > 4.0 m/s or/and aortic valve area (AVA) < 1cm2 or/and AVA indexed to body surface area (BSA) of <0.6 cm2/m2.
* Patients are considered at high risk for mortality with conventional surgical aortic valve replacement as assessed by a Heart Team consisting of at least a cardiologist and surgeon.
* Patients with anatomic characteristics suitable for TAVI based on the local Heart Team decision.
* Patients receiving beta-blockers as a part of their indicated treatment plan.
* Patient understands the purpose, the potential risks as well as benefits of the trial and is willing to participate in all parts of the follow-up.
* Patient has given written consent to participate in the trial.

Exclusion criteria

* A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin, heparin, bivalirudin, clopidogrel, titanium, nickel, cobaltium, chromium, contrast media.
* Patients with permanent pacemaker or defibrillator.
* Ongoing infection, including active endocarditis.
* Echocardiographic evidence of LV or LA thrombus.
* The patient that has any contraindication for antithrombotic treatment.
* Estimated life expectancy of less than 12 months.
* Pregnancy and pre-perimenopause.
* 2nd and 3rd degree atrioventricular (AV) block.
* Bradycardia (<50 beats per minute) at the electrocardiogram (ECG) on the screening/baseline visit.
* Co-morbidity that excludes or significantly interferes with the follow-up visits.
* Enrolment in another study that competes or interferes with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Permanent pacemaker implantation | 7 days
  Permanent pacemaker implantation

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  All-cause mortality
Cardiovascular mortality | 12 months
  Cardiovascular mortality
Shock | 12 months
  Shock necessitating use of inotropic or vasoconstrictive medication
Atrial fibrillation | 12 months
  New documented atrial fibrillation
Ventricular tachycardia/fibrillation | 12 months
  New documented ventricular tachycardia/fibrillation
New conduction abnormalities | 12 months
  complete left bundle branch block, complete right bundle branch block, alternating bundle branch block, 1st grade AV block, 2nd degree AV block, 3rd degree AV block
New severe bradycardia | 12 months
  <50 beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Koliastasis, MD, MSc, Principal Investigator — National and Kapodistrian University of Athens; Odysseas Katsaros, MD, Principal Investigator — National and Kapodistrian University of Athens; Konstantinos Toutouzas, Professor, Study Director — National and Kapodistrian University of Athens
Locations (2):
- Nicosia General Hospital, Nicosia, Cyprus
- First Department of Cardiology, National and Kapodistrian University of Athens, Athens, Attica, Greece

REFERENCES:
- [Background] Aurigemma G, Battista S, Orsinelli D, Sweeney A, Pape L, Cuenoud H. Abnormal left ventricular intracavitary flow acceleration in patients undergoing aortic valve replacement for aortic stenosis. A marker for high postoperative morbidity and mortality. Circulation. 1992 Sep;86(3):926-36. doi: 10.1161/01.cir.86.3.926. PMID 1516206
- [Background] Authors/Task Force members; Elliott PM, Anastasakis A, Borger MA, Borggrefe M, Cecchi F, Charron P, Hagege AA, Lafont A, Limongelli G, Mahrholdt H, McKenna WJ, Mogensen J, Nihoyannopoulos P, Nistri S, Pieper PG, Pieske B, Rapezzi C, Rutten FH, Tillmanns C, Watkins H. 2014 ESC Guidelines on diagnosis and management of hypertrophic cardiomyopathy: the Task Force for the Diagnosis and Management of Hypertrophic Cardiomyopathy of the European Society of Cardiology (ESC). Eur Heart J. 2014 Oct 14;35(39):2733-79. doi: 10.1093/eurheartj/ehu284. Epub 2014 Aug 29. No abstract available. PMID 25173338
- [Background] Brugada J, Katritsis DG, Arbelo E, Arribas F, Bax JJ, Blomstrom-Lundqvist C, Calkins H, Corrado D, Deftereos SG, Diller GP, Gomez-Doblas JJ, Gorenek B, Grace A, Ho SY, Kaski JC, Kuck KH, Lambiase PD, Sacher F, Sarquella-Brugada G, Suwalski P, Zaza A; ESC Scientific Document Group. 2019 ESC Guidelines for the management of patients with supraventricular tachycardiaThe Task Force for the management of patients with supraventricular tachycardia of the European Society of Cardiology (ESC). Eur Heart J. 2020 Feb 1;41(5):655-720. doi: 10.1093/eurheartj/ehz467. No abstract available. PMID 31504425
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Lioufas PA, Kelly DN, Brooks KS, Marasco SF. Unexpected suicide left ventricle post-surgical aortic valve replacement requiring veno-arterial extracorporeal membrane oxygenation support despite gold-standard therapy: a case report. Eur Heart J Case Rep. 2022 Feb 2;6(2):ytac020. doi: 10.1093/ehjcr/ytac020. eCollection 2022 Feb. PMID 35233483
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Saito T, Yoshijima N, Hase H, Yashima F, Tsuruta H, Shimizu H, Fukuda K, Naganuma T, Mizutani K, Araki M, Tada N, Yamanaka F, Shirai S, Tabata M, Ueno H, Takagi K, Higashimori A, Watanabe Y, Yamamoto M, Hayashida K. Impact of beta blockers on patients undergoing transcatheter aortic valve replacement: the OCEAN-TAVI registry. Open Heart. 2020 Jul;7(2):e001269. doi: 10.1136/openhrt-2020-001269. PMID 32641381
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur J Cardiothorac Surg. 2021 Oct 22;60(4):727-800. doi: 10.1093/ejcts/ezab389. No abstract available. PMID 34453161
- [Background] Younis A, Orvin K, Nof E, Barabash IM, Segev A, Berkovitch A, Guetta V, Assali A, Kornowski R, Beinart R. The effect of periprocedural beta blocker withdrawal on arrhythmic risk following transcatheter aortic valve replacement. Catheter Cardiovasc Interv. 2019 Jun 1;93(7):1361-1366. doi: 10.1002/ccd.28017. Epub 2018 Nov 29. PMID 30489692
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572
- [Derived] Koliastasis L, Kim WK, Toutouzas K. Pacemaker Implantation After TAVR: Searching for the Golden Ratio. JACC Cardiovasc Interv. 2023 Aug 14;16(15):1946. doi: 10.1016/j.jcin.2023.06.002. No abstract available. PMID 37587606